CLINICAL TRIAL: NCT01635738
Title: Probiotics and Allergic Diseases
Acronym: probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GenMont Biotech Incorporation (Industry)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TH-IRB-10-14
Record Dates: First submitted 2012-07-04; First posted 2012-07-10 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Atopic Dermatitis; Asthma
Keywords: Probiotics; Lactobacillus paracasei GMNL-133; Lactobacillus fermentum GM-090; Atopic dermatitis; Asthma; Lactobacillus paracasei; Lactobacillus fermentum; efficacy and safety
MeSH Terms: conditions — Dermatitis, Atopic; Asthma

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LP GMNL-133 group (Experimental): Arm: LP GMNL-133 group One capsule with 2x10^9 (cfu) LP GMNL-133, once daily, PO
  Interventions: Biological: LP GMNL-133 capsule
- LF GM-090 group (Experimental): Arm: LF GM-090 group One capsule with 2x10^9 (cfu) LF GM-090, once daily, PO
  Interventions: Biological: LF GM-090 capsule
- LP GMNL-133+LF GM-090 group (Experimental): One capsule with 2x10^9 (cfu) LP GMNL-133+ 2x10^9 (cfu)LF GM-090, once daily, PO
  Interventions: Biological: LP GMNL-133 +LF GM-090 capsule
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: LP GMNL-133 capsule — One capsule with 2x10^9 (cfu) LP GMNL-133, once daily, PO
  Arms: LP GMNL-133 group
Biological: LF GM-090 capsule — Arm: LF GM-090 group One capsule with 2x10^9 (cfu) LF GM-090, once daily, PO
  Arms: LF GM-090 group
Biological: LP GMNL-133 +LF GM-090 capsule — One capsule with 4x10^9 (cfu) LP GMNL-133 +LF GM-090, once daily, PO
  Arms: LP GMNL-133+LF GM-090 group
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Many studies had demonstrated that probiotics could be applied in the prevention and adjuvant treatment for allergic diseases. In this study, we investigate the effects of Lactobacillus paracasei GMNL-133(LP), Lactobacillus fermentum GM-090 (LF), and Lactobacillus paracasei GMNL-133(LP) with Lactobacillus fermentum GM-090 (LF) combination products used for adjuvant treatment of atopic dermatitis and asthma.

DETAILED DESCRIPTION:
The main purpose: To investigate if Lactobacillus paracasei GMNL-133(LP), Lactobacillus fermentum GM-090(LF), Lactobacillus paracasei GMNL-133 (LP) with Lactobacillus fermentum GM-090 (LF) combination products could be used for the adjuvant treatment of atopic dermatitis and asthma.

The Secondary Objective: To investigate whether probiotics consumption improve the quality of life and allergic symptoms to different people with Lactobacillus paracasei GMNL-133 (LP), Lactobacillus fermentum GM-090 (LF) and Lactobacillus paracasei GMNL-133(LP) and Lactobacillus fermentum GM-090 (LF) combination products.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 1 year old and 18 years old,
2. AD cases fulfill the diagnostic criteria by Hannifin and Rajka.
3. Atopy as shown by at least one positive skin test (weal size ≧ 3mm) or one positive MAST (RAST) (IgE ≧ 0.7 kU/L) test to any common food or environmental allergens.

Exclusion Criteria:

1. Systematic corticosteroid, immunosuppressive therapy, or antimycotics treatment during the 4 weeks, antihistamines, and singulair during the 7 days before enrollment
2. Probiotic preparations used within 2 weeks before entering the study
3. Use of antibiotics now or other oral medications that will interfere the results
4. If they had immune deficiency disease or other major medical problems
5. If they had participated in another clinical study during the past month.
6. Subjects are undergoing desensitization therapy within 3 months prior to the screening period.
7. Subjects have participated investigational drug trial within 4 weeks before entering this study.
8. Subjects are pregnant, lactating or planning to become pregnant.
9. Subjects with any other serious diseases considered by the investigator that could interfere with the performance of SCORAD score result.
10. Subjects who is lack of physical integrity of gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The Effects of probiotics in improving life quality and symptomatic severity | 2 years
  1. Atopic dermatitis
     Primary Endpoints:
     SCORAD score, Children's Dermatology Life Quality Index (CDLQI), and Dermatitis Family Impact Questionnaire
  2. Asthma
     Primary Endpoints:
     GINA guideline asthma severity ( step up or step down) ACT, PAQLQ, PACQLQ, PASS Questionnaire
  3. Allergic Rhinitis
  Primary Endpoints:
  ARIA allergic rhinitis severity PRQLQ, NTSS Questionnaire

SECONDARY OUTCOMES:
The Effects of probiotics on biomakers and other symptom relief | 2 years
  Atopic dermatitis:
  Decrease topical steroid and oral antihistamine use, changes of skin prick test severity, effect persistency after discontinuing Lactobacillus paracasei GMNL-133, Lactobacillus fermentum GM-090 or the composition of Lactobacillus paracasei GMNL-133 and Lactobacillus fermentum GM-090 intake, changes of cytokine and IgE, urine EPX, 8-ohdg biomarkers.
  Comparison of Probiotic group (LP, LF and LP+LF) and placebo group
  Asthma:
  Peak flow lung function, the changes of skin prick test severity, effect persistency after discontinuing probiotics, ISAAC questionnaire, use of rescue medication, unscheduled visit to emergency unit, changes of cytokine and IgE, urine EPX, 8-ohdg biomarkers Comparison of Probiotic group (LP, LF and LP+LF) and placebo group
  Allergic Rhinitis :
  Changes of skin prick test severity, effect persistency after discontinuing probiotics, ISAAC questionnaire, use of rescue medication, changes of cytokine and IgE, urine EPX, 8-ohdg biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: I-Jen Wang, Doctor, Study Chair — Taipei Hospital, Department of Health, Taiwan, R.O.C.
Locations (1):
- Taipei Hospital, Department of Health, Taiwan, R.O.C., New Taipei City, Taiwan

REFERENCES:
- [Result] Hong HJ, Kim E, Cho D, Kim TS. Differential suppression of heat-killed lactobacilli isolated from kimchi, a Korean traditional food, on airway hyper-responsiveness in mice. J Clin Immunol. 2010 May;30(3):449-58. doi: 10.1007/s10875-010-9375-8. Epub 2010 Mar 5. PMID 20204477
- [Result] Yao TC, Chang CJ, Hsu YH, Huang JL. Probiotics for allergic diseases: realities and myths. Pediatr Allergy Immunol. 2010 Sep;21(6):900-19. doi: 10.1111/j.1399-3038.2009.00955.x. Epub 2009 Dec 9. PMID 20003066
- [Result] Park CW, Youn M, Jung YM, Kim H, Jeong Y, Lee HK, Kim HO, Lee I, Lee SW, Kang KH, Park YH. New functional probiotic Lactobacillus sakei probio 65 alleviates atopic symptoms in the mouse. J Med Food. 2008 Sep;11(3):405-12. doi: 10.1089/jmf.2007.0144. PMID 18800885
- [Result] Peng GC, Hsu CH. The efficacy and safety of heat-killed Lactobacillus paracasei for treatment of perennial allergic rhinitis induced by house-dust mite. Pediatr Allergy Immunol. 2005 Aug;16(5):433-8. doi: 10.1111/j.1399-3038.2005.00284.x. PMID 16101937
- [Result] Wang MF, Lin HC, Wang YY, Hsu CH. Treatment of perennial allergic rhinitis with lactic acid bacteria. Pediatr Allergy Immunol. 2004 Apr;15(2):152-8. doi: 10.1111/j.1399-3038.2004.00156.x. PMID 15059192
- [Derived] Wang IJ, Wang JY. Children with atopic dermatitis show clinical improvement after Lactobacillus exposure. Clin Exp Allergy. 2015 Apr;45(4):779-87. doi: 10.1111/cea.12489. PMID 25600169